CLINICAL TRIAL: NCT06682065
Title: Telemedicine Contraceptive Counselling (TECC) Versus Standard Care - a Pilot and Randomized Controlled Trial of Periabortion Contraceptive Counseling
Brief Title: Telemedicine Contraceptive Counselling (TECC) Versus Standard Care
Acronym: TECC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: University of Cape Town (Other)
Responsible Party: Principal Investigator, Margit Endler, Associate Professor, MD ObGyn, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: TECC
Record Dates: First submitted 2024-04-08; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Contraceptive Usage; Telemedicine
MeSH Terms: conditions — Contraception Behavior | interventions — Telemedicine; Standard of Care

STUDY DESIGN:
Intervention Model Description: 1:1
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemedicine (Experimental): WhatsApp algorithmic chatbot see further description
  Interventions: Other: Telemedicine for contraceptive counseling (TECC)
- Standard Care (Active Comparator): Standard of care contraceptive counseling with clinic nurse
  Interventions: Other: Standard Care

INTERVENTIONS:
Other: Telemedicine for contraceptive counseling (TECC) — WhatsApp algorithmic chatbot that screens preferences and medical eligibility to recommend two methods, informs about all methods, allows choice out of all methods, produce summary to substitute for clinical record
  Arms: Telemedicine
Other: Standard Care — In-personcontraceptive counseling with a nurese according to clinical standard of care
  Arms: Standard Care

SUMMARY:
Overall purpose of the PILOT and RCT:

This research project aims to increase access and uptake of contraception after abortion through the systematic development and testing of a new telemedicine service for contraceptive counselling (TECC). The investigators will perform a pilot study in South Africa, and multicenter randomized controlled trial in South Africa and Kenya with the following specific aims:

DETAILED DESCRIPTION:
Overall purpose of the PILOT and RCT:

This research project aims to increase access and uptake of contraception after abortion through the systematic development and testing of a new telemedicine service for contraceptive counselling (TECC). The investigators will perform a pilot study in South Africa, and multicenter randomized controlled trial in South Africa and Kenya with the following specific aims:

1. To design and test a user-friendly online service for contraceptive counseling informed by systematic research into the preference and experience of women in our study setting.
2. To compare uptake of long-acting reversible contraception (LARC) after TECC and in-person contraceptive counseling.
3. To compare rates of choice, uptake, and continuation of LARC or any contraceptive, satisfaction, preference for counseling, recurrent unintended pregnancy, and recurrent abortion after TECC and in-person contraceptive counseling.

PILOT STUDY Objective: To assess the acceptability of a new online e-health service for contraceptive counselling i.e., telemedicine contraceptive counseling (TECC)

Design: A mixed methods pilot study developing and testing a new TECC service preceding a randomized controlled trial Setting and duration: The study will take place at Mitchell's Plain's community health center (CHC) in Western Cape, between February November 2023 and December 2023.

Study population: 30 women seeking abortion either medical or surgical, ≥ 18 years of age, able to communicate and understand spoken and written English, with private access to a smartphone, and willing to participate in the study

Recruitment and consent: Recruitment, informed consent, baseline interview and randomization will take place at the clinics by one of two experienced field workers, fluent in English and isiXhosa/Afrikaans.

Intervention: Participants will test the TECC service while waiting at the clinic to see the nurse for their abortion consultation. A follow-up survey will be sent out and completed by phone if necessary at 2 weeks after enrolment in the study. Out of these 30 women, approximately 10 (or until data saturation is achieved) will participate in semi-structured in-depth interviews regarding their experience of using the TECC service.

Primary outcome collected at 2 weeks Main outcome variable will be a compound variable reflecting the proportion of women who choose a method after completing the TECC intervention and report 1) being satisfied or very satisfied with the service (affective attitude), 2) understanding the content and purpose of the intervention (coherence), 3) feeling confident in their ability to use the service (self-efficacy), 4) experiencing the service as easy to use (burden), 5) assessing service as likely to be of use in the community (effectiveness)

Secondary outcomes collected at 2 weeks

1. Contraceptive method chosen by type (%)
2. Choice of LARC (%), defined as choice of an IUD or a subdermal implant for contraception
3. Change of method with respect to previous use (%)

Qualitative component Data collection - qualitative component Data will be collected through semi structured in depth interviews (IDIs), held in person or by phone after the second quantitative data collection point. The sample size is estimated to be until data saturation or up to 10 interviews. The interview guide for the IDIs will be developed to capture measures of the acceptability of the TECC service according to Sekhon et al.'s framework, i.e. how participants feel about the intervention (affective attitude), how much effort is required to participate in the intervention (burden), how well the intervention fits with the participants value system (ethicality), how well the intervention is understood (coherence), what benefits must be given up to utilize the intervention (opportunity costs), how likely the intervention is to work (perceived effectiveness), and the participants confidence in being able to use the intervention (self-efficacy). Emphasis will be on enhancing the quantitative findings and gaining a more comprehensive understanding of the acceptability of the TECC intervention. Especially aspects of the framework that are more difficult to explore quantitatively, such as ethicality and opportunity costs will be explored. Questions will be open ended, allowing new themes to emerge from the data, and the interview guide may be adapted to accommodate and explore themes emerging in the interviews.

RANDOMIZED CONTROLLED TRIAL

Objective:

Setting:

Population: 510 women seeking abortion either medical or surgical, < 13+0 weeks gestation, ≥18 years of age, able to communicate and understand spoken and written English, with private access to a smart phone, and willing to participate in the study.

Recruitment and consent: Recruitment, informed consent, baseline interview and randomization will take place at the clinics by one of two experienced field workers, fluent in English and isiXhosa/Afrikaans.

RCT: Participants will be randomly assigned to either standard care or TECC.

1. Standard care: Contraceptive counselling with clinic nurse.
2. TECC: While waiting for their abortion consultation with the clinic nurse, participants will use their phones to complete a contraceptive counseling session through the TECC service.

Outcome measures: The investigators will compare effectiveness and acceptability of the service between the telemedicine and the standard care arm. Follow-up will through links ot online surveys in RedCap at 12 weeks, 6 months and 12 months after the initial consultation.

Primary outcome at 12 weeks Uptake of LARC, defined as uptake of an IUD or a subdermal implant for contraception, within 12 weeks Secondary outcomes at 12 weeks

1. choice of LARC
2. uptake of any contraception
3. choice or uptake of new method with regards to previous use
4. satisfaction with TECC service (using a a multi-question validated scale)
5. Rated use of service for decision making (using a multi-question validated scale)
6. Degree of agency in decision making (using a a multi-question validated scale)
7. preference for counselling Secondary outcomes at 6 months

1. continued use of LARC 2. continued use of any contraception 3. recurrent unintended pregnancy 4. recurrent abortion Secondary outcomes at 12 months

1. continued use of LARC
2. continued use of any contraception
3. recurrent unintended pregnancy
4. recurrent abortion
5. Change of method at any timepoint up to 12 months
6. Reason for change of method

ELIGIBILITY:
* Seeking either surgical or medical abortion
* ≥ 18 years of age
* Able to communicate and understand spoken and written English
* With private access to a smart phone
* Willing to participate in the study procedures

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 510 (Estimated)
Dates: Start 2024-05-05 (Actual); Primary Completion 2025-02-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Use of LARC (IUD or progestin implant) at 12 week follow-up | 12 weeks
  Proportion of participants in each arm with using LARC (IUD or progestin implant) at 12 week follow-up

SECONDARY OUTCOMES:
Choice of LARC on day of consultation | Baseline
  Proportion of participants in each arm chosing LARC on day of first visit (recruitment)
Use of LARC at 6 months | 6 months
  Proportion of participants in each arm using LARC at 6 months follow-up
Use of LARC at 12 months | 12 months
  Proportion of participants in each arm using LARC at 12 months follow-up
Unplanned pregnancy within 6 months | 6 months
  Proportion of participants in each arm with unplanned pregnancy recorded at 6 month follow-up and having occurred since previous abortion
Unplanned pregnancy within 12 months | 12 months
  Proportion of participants in each arm with unplanned pregnancy recorded at 12 month follow-up and having occurred since previous abortion.
Recurrent abortion within 6 months | 6 months
  Proportion of participants in each arm with recurrent abortion recorded at 6 month follow-up and having occurred since previous abortion
Recurrent abortion within 12 months | 12 months
  Proportion of participants in each arm with recurrent abortion recorded at 12 month follow-up and having occurred since previous abortion
Preference for counseling model | Baseline
  Proportion of participants in each arm using expressing preference for telemedicine counseling model
Satisfaction with contraceptive counseling | Baseline
  validated scale (0-6)
Decision-competence after contraceptive counseling | Baseline
  validated scale (0-100)
Agency in contraceptive decision making | Baseline
  modified validated scale
Change of contraceptive method | 12 months
  Change of contraceptive method

CONTACTS AND LOCATIONS:
Overall Officials: Margit Endler, PhD, Principal Investigator — Karolinska Institutet
Locations (2):
- South Africa (2):
  - Michael Mapongwana, Cape Town
  - Mitchell´s Plain CHC, Cape Town

IPD SHARING:
Plan to Share IPD: No
Pseudonymized data will be made available to other researchers upon reasonable request

DOCUMENTS (1):
  • Study Protocol (2024-04-08): https://cdn.clinicaltrials.gov/large-docs/65/NCT06682065/Prot_000.pdf